CLINICAL TRIAL: NCT05740280
Title: iCP-NI - A Phase 1, Double Blind, Placebo Controlled, Single and Multiple Intravenous Infusion, Safety, Tolerability, Pharmacokinetic, and Immunogenicity Study in Healthy Male and Female Subjects
Brief Title: iCP-NI - Safety, Tolerability, Pharmacokinetic, and Immunogenicity Study in Healthy Male and Female Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed by Sponsor for business reasons
Sponsor: Cellivery Therapeutics, Inc. (Industry)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CV_iCP-NI_002
Record Dates: First submitted 2023-02-05; First posted 2023-02-23 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
Keywords: COVID-19; Pneumonia; Virus Diseases; Infections
MeSH Terms: conditions — COVID-19; Pneumonia; Virus Diseases; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- iCP-NI (Experimental): Part A will comprise a single dose, sequential group design. Part A: 40 subjects will be studied in 5 groups (Groups A1 to A5). In each of Groups A1 to A5, 6 subjects will receive iCP-NI and 2 subjects will receive placebo.
  Part A: Five proposed dose levels per protocol.
  Part B will comprise a multiple dose, sequential group design. Part B: 24 subjects will be studied in 3 groups (Groups B1 to B3). In each of Groups B1 to B3, 6 subjects will receive iCP-NI and 2 subjects will receive placebo.
  Part B: Proposed dose levels to be determined following review of available data from Part A.
  Interventions: Drug: iCP-NI
- Placebo (Placebo Comparator): Part A will comprise a single dose, sequential group design. Part A: 40 subjects will be studied in 5 groups (Groups A1 to A5). In each of Groups A1 to A5, 6 subjects will receive iCP-NI and 2 subjects will receive placebo.
  Part A: Five proposed dose levels per protocol.
  Part B will comprise a multiple dose, sequential group design. Part B: 24 subjects will be studied in 3 groups (Groups B1 to B3). In each of Groups B1 to B3, 6 subjects will receive iCP-NI and 2 subjects will receive placebo.
  Part B: Proposed dose levels to be determined following review of available data from Part A.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: iCP-NI — 20 mg/mL iCP-NI solution for intravenous injection
  Arms: iCP-NI
Drug: Placebo — Placebo solution for intravenous injection
  Arms: Placebo

SUMMARY:
This is a Phase 1, double-blind, randomized, placebo-controlled study to investigate single and multiple intravenous infusions of improved cell-permeable nuclear import inhibitor (iCP NI) in healthy subjects.

DETAILED DESCRIPTION:
Improved cell-permeable nuclear import inhibitor (iCP-NI) is a synthetically manufactured, cell-penetrating peptide which has been developed by fusion of advanced macromolecule transduction domain of hydrophobic cell-permeable peptide and nuclear factor kappa-light- chain-enhancer of activated B cells (NF-κB)-derived nuclear localization sequence.

The production and secretion of cytokines from innate immune cells are critical responses to inflammation and infection in the body.

iCP-NI is a binding competitor that inhibits the interaction of nuclear transfer material proteins such as IATF (NF-BB, STAT, AP-1, NFAT) and importin alpha5, inhibiting the nuclear transport of IATF to prevent inflammatory cytokine transcription.

This study is the first-human clinical trial for iCP-NI which is intended to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of iCP-NI.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all of the following criteria at the screening visit unless otherwise stated:

* Males or females, of any race, between 18 and 55 years of age, inclusive.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is acceptable) at screening and check in, from the physical examination performed between screening and check-in, and from the 12-lead ECG and vital signs measurements performed at screening, as assessed by the investigator (or designee).
* Females of nonchildbearing potential, defined as permanently sterile (ie, due to hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or Mullerian agenesis) or postmenopausal. Females will not be pregnant or lactating. Males will agree to use contraception.
* Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.

Exclusion Criteria:

Medical conditions

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
* Any of the following:

  1. QTcF >450 ms in males or >470 ms in females, confirmed by calculating the mean of the original value and 2 repeats.
  2. QRS duration >110 ms, confirmed by calculating the mean of the original value and 2 repeats
  3. PR interval >220 ms, confirmed by calculating the mean of the original value and 2 repeats.
  4. findings that would make QTc measurements difficult or QTc data uninterpretable.
  5. history of additional risk factors for torsades de pointes (eg, heart failure, hypokalemia, family history of long QT syndrome).
* Confirmed (eg, 2 consecutive measurements) systolic blood pressure >140 or <90 mmHg, diastolic blood pressure >90 or <50 mmHg, and pulse rate >100 or <40 beats per minute.
* Positive hepatitis panel and/or positive human immunodeficiency virus test. Subjects whose results are compatible with prior immunization may be included at the discretion of the investigator.
* Absolute neutrophil count, absolute lymphocyte count, or white blood cell count that is below the institution's lower limit of normal.

Prior/concomitant therapy

* Administration of a COVID 19 vaccine in the 30 days prior to dosing.
* Use or intend to use any prescription medications/products within 14 days prior to dosing, unless deemed acceptable by the investigator (or designee).
* Use or intend to use slow release medications/products considered to still be active within 14 days prior to check in, unless deemed acceptable by the investigator (or designee).
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 7 days prior to check in, unless deemed acceptable by the investigator (or designee).

Prior/concurrent clinical study experience

* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days (or 5 half-lives, whichever is longer) prior to dosing.
* Have previously completed or withdrawn from this study or any other study investigating iCP-NI, and have previously received iCP-NI.

Diet and lifestyle

* Alcohol consumption of >21 units per week for males and >14 units per week for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
* Positive urine drug screen at screening or check-in or positive alcohol urine or breath test result at check in.
* History of alcoholism or drug/chemical abuse within 2 years prior to check in.
* Use of tobacco or nicotine containing products within 3 months prior to check in.
* Ingestion of poppy seed containing foods or beverages within 7 days prior to check-in.

Other exclusions

* Receipt of blood products within 2 months prior to check in.
* Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
* Poor peripheral venous access.
* Subjects who, in the opinion of the investigator (or designee), should not participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Part A: Incidence and severity of adverse events (AEs) | Screening to Follow Up (Day 28+2 days)
Part B: Incidence and severity of adverse events (AEs) | Screening to Follow Up (Day 28+2 days)
Part A: Incidence of laboratory abnormalities, based on hematology, clinical chemistry, and urinalysis test results | Screening to Follow Up (Day 7)
Part B: Incidence of laboratory abnormalities, based on hematology, clinical chemistry, and urinalysis test results | Screening to Follow Up (Day 28+2 days)
Part A: Number of participants with abnormal 12-lead ECG parameters | Screening to Follow Up (Day 7)
Part B: Number of participants with abnormal 12-lead ECG parameters | Screening to Follow Up (Day 28+2 days)
Part A: Number of participants with abnormal vital signs measurements | Screening to Follow Up (Day 7)
Part B: Number of participants with abnormal vital signs measurements | Screening to Follow Up (Day 28+2 days)
Part A: Number of participants with abnormal physical examinations | Screening to Follow Up (Day 7)
Part B: Number of participants with abnormal physical examinations | Screening to Follow Up (Day 28+2 days)

SECONDARY OUTCOMES:
Part A: Pharmacokinetics (PK): Area under the concentration time curve from time 0 extrapolated to infinity (AUC0-∞) of iCP-NI | Day 1: Pre-dose up to 12 hours post start of infusion
Part B: Pharmacokinetics (PK): Area under the concentration time curve from time 0 extrapolated to infinity (AUC0-∞) of iCP-NI | Day 1 (Pre-dose) up to Day 7 (12 hours post start of infusion)
Part A: Pharmacokinetics (PK): Area under the concentration time curve from time 0 to the time of the last quantifiable concentration (AUC0-tlast) of iCP-NI | Day 1: Pre-dose up to 12 hours post start of infusion
Part B: Pharmacokinetics (PK): Area under the concentration time curve from time 0 to the time of the last quantifiable concentration (AUC0-tlast) of iCP-NI | Day 1 (Pre-dose) up to Day 7 (12 hours post start of infusion)
Part A: Pharmacokinetics (PK): Area under the concentration-time curve over a dosing interval (τ) (AUC0-τ) of iCP-NI | Day 1: Pre-dose up to 12 hours post start of infusion
Part B: Pharmacokinetics (PK): Area under the concentration-time curve over a dosing interval (τ) (AUC0-τ) of iCP-NI | Day 1 (Pre-dose) up to Day 7 (12 hours post start of infusion)
Part A: Pharmacokinetics (PK): Maximum observed concentration (Cmax) of iCP-NI | Day 1: Pre-dose up to 12 hours post start of infusion
Part B: Pharmacokinetics (PK): Maximum observed concentration (Cmax) of iCP-NI | Day 1 (Pre-dose) up to Day 7 (12 hours post start of infusion)
Part A: Pharmacokinetics (PK): Time of the maximum observed concentration (tmax) of iCP-NI | Day 1: Pre-dose up to 12 hours post start of infusion
Part B: Pharmacokinetics (PK): Time of the maximum observed concentration (tmax) of iCP-NI | Day 1 (pre-dose) up to Day 7 (12 hours post start of infusion)
Part A: Pharmacokinetics (PK): Apparent terminal elimination half life (t1/2) of iCP-NI | Day 1: Pre-dose up to 12 hours post start of infusion
Part B: Pharmacokinetics (PK): Apparent terminal elimination half life (t1/2) of iCP-NI | Day 1 (Pre-dose) up to Day 7 (12 hours post start of infusion)
Part A: Pharmacokinetics (PK): Accumulation ratio based on AUC0-τ (ARAUC) of iCP-NI | Day 1: Pre-dose up to 12 hours post start of infusion
Part B: Pharmacokinetics (PK): Accumulation ratio based on AUC0-τ (ARAUC) of iCP-NI | Day 1 (Pre-dose) up to Day 7 (12 hours post start of infusion)
Part A: Serum concentrations of anti-iCP-NI antibodies | Day -1, Follow up (Day 7) and Immunogenicity Visit (Day 28 + 2 days)
  Serum concentrations of anti-iCP-NI antibodies will be determined using a validated analytical procedure.
Part B: Serum concentrations of anti-iCP-NI antibodies | Day -1, Day 7 (pre-am dose) and Follow up (Day 28 + 2 days)
  Serum concentrations of anti-iCP-NI antibodies will be determined using a validated analytical procedure.
Part A: Serum concentrations of neutralizing antibodies | Day -1, Follow up (Day 7) and Immunogenicity Visit (Day 28 + 2 days)
  Serum concentrations of neutralizing antibodies will be determined using a validated analytical procedure.
Part B: Serum concentrations of neutralizing antibodies | Day -1, Day 7 (pre-am dose) and Follow up (Day 28 + 2 days)
  Serum concentrations of neutralizing antibodies will be determined using a validated analytical procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Clinical Research Unit Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided